CLINICAL TRIAL: NCT05341362
Title: Hemodynamic Management Target on Continuous Monitoring in Cesarean Delivery-A Randomized Controlled Trial in Patients With Supine Hypotensive Syndrome
Brief Title: Hemodynamic Management in Women With SHS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University, China (Other)
Responsible Party: Principal Investigator, Yuqing Li, Undergraduate doctor, China Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SHSandLidco
Record Dates: First submitted 2022-04-10; First posted 2022-04-22 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Supine Hypotensive Syndrome
Keywords: supine hypotensive syndrome; cesarean delivery; spinal anesthesia; CSEA

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blank Group (No Intervention): In this group, the anesthesia management is conducted according to the anesthetists' experience, based on the regular monitor.
- LiDCOrapid Group (Experimental): In this group, the anesthesia management is conducted based on both the regular monitor and the hemodynamic figures on the LiDCOrapid.
  Interventions: Procedure: LiDCOrapid

INTERVENTIONS:
Procedure: LiDCOrapid — According to the illustration of the patient's hemodynamic figures shown on the LiDCOrapid monitor, we decide on the timing of the vasopressor administration. This group aims to maintain the cardiac output within a baseline range.
  Arms: LiDCOrapid Group

SUMMARY:
Supine hypotensive syndrome often occurs following spinal anesthesia for cesarean delivery.In our study we base the regulation and drug administration both on the regular monitor and on a novel monitor which reflects upon the hemodynamic changes. Our aim is to observe whether the outcome of SHS patients with anesthesia management based on hemodynamic figures differs from those based on experience.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) Physical Status Classification II and had no significant cardiovascular, pulmonary, renal or endocrine disease, without contraindications to CSEA,and could be diagnosed as SHS according to the criteria.

Exclusion Criteria:

* Patients undergoing emergency CD, CD under general anesthesia or patients' refusal to participate, or multiple fetations.

Ages: 22 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — The disease supine hypotensive syndrome happens among pregnant women in their late pregnancy. Therefore, the participants should be female.
Enrollment: 60 (Estimated)
Dates: Start 2022-04-17 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Umbilical arterial blood gas PH | 30minutes
  The value is tested immediately after the blood sample is achieved after the infant is born.

SECONDARY OUTCOMES:
Discomfort Score | 1day
  we explored a scoring system to quantify the SHS symptom scale from 0 to 8, score high means more symptoms of SHS occurred
total vasopressor dosage | 30 minutes
  total vasopressor given during the time span between the operation began to the baby was delivered
Umbilical blood gas lactate | 30minutes
  The value is tested immediately after the blood sample is achieved after the infant is born.
Time span | 2 hours
  the period between the operation began to the baby was delivered

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Undecided